CLINICAL TRIAL: NCT04981145
Title: The Efficacy and Safety of Iguratimod (IGU) in the Treatment of Primary Sjögren's Syndrome: a Multi-center, Prospective, Open Study
Brief Title: The Efficacy and Safety of Iguratimod (IGU) in the Treatment of Primary Sjögren's Syndrome
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0391
Record Dates: First submitted 2021-07-05; First posted 2021-07-28 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Primary Sjögren's Syndrome
Keywords: Primary Sjögren's syndrome; Sjögren's syndrome; Iguratimod
MeSH Terms: conditions — Sjogren's Syndrome | interventions — iguratimod; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IGU Group (Experimental)
  Interventions: Drug: Iguratimod Tablets
- HCQ Group (Active Comparator)
  Interventions: Drug: Hydroxychloroquine Sulfate Tablets

INTERVENTIONS:
Drug: Iguratimod Tablets — Participants are treated with Iguratimod Tablets 25 mg Twice a day for 24 weeks.
  Arms: IGU Group
Drug: Hydroxychloroquine Sulfate Tablets — Participants are treated with Hydroxychloroquine Sulfate Tablets 200 mg Twice a day for 24 weeks.
  Arms: HCQ Group

SUMMARY:
A multi-center, prospective, open-label, randomized controlled study of efficacy and safety of Iguratimod in patients with Primary Sjögren's syndrome

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with pSS by meeting the 2016 ACR/EULAR Classification Criteria.
* The patient complained of dry mouth and eyes.
* Positive anti-SSA/Ro-60 antibody at screening.
* IgG≥16 g/L.
* No hormone, immunosuppressant, biological agents or other treatments were received within 4 weeks before screening;
* Pregnancy test of is negative. Use effective contraceptives during the trial (female)
* Those who did not participate in any drug trial within 12 weeks before enrollment

Exclusion Criteria:

* Pregnant or lactating or planning to get pregnant during the duration of the study.
* Complicated with other CTD
* Complicated with malignancy
* mental illness, a history of alcohol abuse, immunodeficiency, uncontrolled infections, and drug or other substance abuse
* serious systemic damage, glucocorticoids, other immunosuppressants and biological agents should be added to control the condition: Heart, liver (transaminase/bilirubin >1.5 times the upper normal limit), kidney (Cr≥133mmol/L), lung (FVC % < 60%), blood (white blood cell <3×109/L, HGB<80g/L, PLT<80×109/L), etc.
* Fundus/visual field lesions;
* Allergic to any component of the study drug (IGU and/or HCQ);
* the investigator considers the patient to be unsuitable for entry into the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The change of SSRI-30 between the two groups at 24 weeks | 24 weeks
  SS Responder Index (SSRI) is a composite endpoint, investigators defined an SSRI-30 response as a ≥30% improvement in at least two of five outcome measures (patient-assessed visual analogue scale scores for fatigue, oral dryness and ocular dryness, unstimulated whole salivary flow and ESR at 24 weeks

SECONDARY OUTCOMES:
Change in The European League Against Rheumatism (EULAR) Sjogren's Syndrome Patient Reported Index (ESSPRI) score from Baseline to Week 24 | 24 weeks
  The ESSPRI is composed of 3 scales - dryness, fatigue, and pain. Each scale is measured 0 - 10, 0 being no symptoms, 10 being maximal imaginable dryness, fatigue or pain. The total score is the mean score of the three scales. Baseline ESSPRI total score will be compared to week 24, end of treatment, ESSPRI total score.
Change in total score of the EULAR Sjogren's syndrome disease activity index (ESSDAI) from baseline to week 24 | 24 weeks
  The ESSDAI is a disease activity measurement that has 12 domains. The score of each domain is the product of the weight of the domain by the level of activity. Activity levels are 0 - 3, 0 being no activity, 3 being high activity. The total score is the sum of the score of all domains. Change in total score from BL to week 24 will be measured.
Change in Schimer's test | 24 weeks
  The change from baseline in Schimer's test at 24 weeks. The Schirmer's test assesses tear secretion.
Change in Immunoglobulin G (IgG) concentration | 10 and 24 weeks
  The change from baseline in IgG concentration at 10 and 24 weeks.
Change in serum complements C3 and C4 concentration | 10 and 24 weeks
  The change from baseline in serum complements C3 and C4 concentrationat 10 and 24 weeks.
Change in titer of Rheumatoid Factors | 10 and 24 weeks
  The change from baseline in titer of rheumatoid factors at 10 and 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Yongmei Han, Principal Investigator — Sir Run Run Shaw Hospital; Hongzhi Wang, Principal Investigator — Affiliated Hospital of Jiaxing University; Ying Guan, Principal Investigator — Zhuji People's hospital
Locations (1):
- Second affiliated hospital of zhejiang university，school of medical, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen X, Zhang T, Meng L, Xu C, Jiang L, Wang G, Hou T, Wang H, Han Y, Guan Y, Wang Y, Xue J. Efficacy and safety of iguratimod in patients with primary Sjogren's syndrome: a multicentre randomised controlled trial. RMD Open. 2025 Dec 21;11(4):e006180. doi: 10.1136/rmdopen-2025-006180. PMID 41423293